CLINICAL TRIAL: NCT05024812
Title: An Open Label, Single Arm, Multicenter Phase Ⅰb/Ⅱ Clinical Study of Fruquintinib Combined With Toripalimab and SOX Regimen in the First-line Treatment of Advanced Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: Fruquintinib Combined With Toripalimab and SOX Regimen in the First-line Treatment of Advanced Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Feng Wang, Professor, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-013-FLAG-G102
Record Dates: First submitted 2021-08-20; First posted 2021-08-27 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Metastatic Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): fruquintinib + toripalimab + SOX
  Interventions: Drug: fruquintinib＋toripalimab + SOX

INTERVENTIONS:
Drug: fruquintinib＋toripalimab + SOX — phase Ib: fruquintinib (dose finding): L1: 3 mg/d，L2: 4 mg/d，L3: 5 mg/d, qd po, D1-14, Q3W toripalimab: 240mg, I.V., D1, Q3W; S-1: 40-60mg bid, D1-14, Q3W; Oxaliplatin: 130mg/m^2, ivgtt 2h, D1,Q3W. phase II: fruquintinib: RP2D toripalimab: 240mg, I.V., D1, Q3W; S-1: 40-60mg bid, D1-14, Q3W; Oxaliplatin: 130mg/m^2, ivgtt 2h, D1,Q3W.

SUMMARY:
This is a prospective, open-label, multicenter, single arm phase Ⅰb/Ⅱ clinical study aims to explore the efficacy and safety of fruquintinib combined with toripalimab and SOX regimen in the first-line treatment of unresectable advanced metastatic gastric or gastroesophageal junction adenocarcinoma.

DETAILED DESCRIPTION:
At present, the first-line standard treatment of metastatic gastric cancer is still doublet or triplet chemotherapy of fluorouracil combined with platinum or paclitaxel. In recent years, immune checkpoint inhibitors (ICIs) have emerged in advanced gastric cancer with their unique mechanism of action. PD-1 monoclonal antibody has been explored in multiple combination schemes in the first-line treatment of advanced gastric cancer. This study aims to explore the efficacy and safety of an antiangiogenetic TKI, fruquintinib combined with an ICI, toripalimab and the standard doublet SOX regimen in the first-line treatment of unresectable advanced metastatic gastric or gastroesophageal junction adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically determined unresectable advanced gastric or gastroesophageal junction adenocarcinoma;
* 18-75 years old (including 18 and 75 years old);
* No previous anti-tumor treatment for metastatic diseases;
* HER2 negative;
* Eastern Cooperation Oncology Group (ECOG) performance status of 0-1;
* Life expectancy ≥ 3 months;
* At least one measurable lesion according to RECIST version 1.1;
* Adequate organ and bone marrow functions:

Absolute neutrophil count≥1.5x10^9/L; Platelet count≥100x10^9/L; Hemoglobin≥9g/dL; Serum bilirubin≤1.5x the upper limit of normal(ULN); Alanine aminotransferase(ALT) and aspartate aminotransferase(AST)≤1.5x ULN; Serum creatinine≤1.5x ULN; Endogenous creatinine clearance rate ≥ 50ml / min;

* Women of childbearing age need to take effective contraceptive measures.

Exclusion Criteria:

* Previous treatment with vascular endothelial growth factor receptor (VEGFR) inhibitors or previous use of immune checkpoint inhibitors;
* Other malignant tumors in the past 5 years, except for skin basal cell or squamous cell carcinoma after radical surgery, or cervical carcinoma in situ;
* There was central nervous system (CNS) metastasis or previous brain metastasis before enrollment;
* Patients with autoimmune diseases or history of autoimmune diseases within 4 weeks before enrollment;
* Previously received allogeneic bone marrow transplantation or organ transplantation;
* Uncontrolled malignant ascites;
* Participated in other unapproved or unlisted drug clinical trials in China within 4 weeks before enrollment, and received corresponding experimental drug treatment;
* Cardiovascular disease, including unstable angina or myocardial infarction, occurred within 6 months before the start of study treatment;
* Subjects allergic to the study drug or any of its adjuvants;
* International normalized ratio (INR) > 1.5 or partially activated prothrombin time (APTT) > 1.5 × ULN；
* The researchers judged clinically significant electrolyte abnormalities;
* At present, the patient has hypertension that cannot be controlled by drugs, which is specified as: systolic blood pressure ≥ 140 mmHg and / or diastolic blood pressure ≥ 90 mmHg;
* Patients currently have poorly controlled diabetes (fasting glucose level is greater than CTCAE grade 2 after regular treatment);
* Patients with dysphagia, active peptic ulcer, intestinal obstruction, active gastrointestinal bleeding, peptic perforation, malabsorption syndrome or uncontrolled intestinal inflammatory diseases;
* Any disease or state affecting drug absorption before enrollment, or the patient cannot take oral medication;
* Patients with obvious evidence of bleeding tendency or medical history within 3 months before enrollment, hemoptysis or thromboembolism within 12 months;
* Cardiovascular diseases with significant clinical significance, including but not limited to acute myocardial infarction, severe / unstable angina pectoris or coronary artery bypass grafting within 6 months before enrollment;
* Ventricular arrhythmia requiring drug treatment;
* Congestive heart failure ≤New York Heart Association (NYHA) class 2;
* LVEF < 50%;
* Active or uncontrolled severe infection ≥ grade 2 according to National Cancer Institute Common Toxicity (NCI-CTC) criteria;
* With positive urine protein and 24-hour urinary protein content>1g;
* Known human immunodeficiency virus (HIV) infection; known history of clinically significant liver disease, including viral hepatitis;
* Pregnant (positive pregnancy test before medication) or lactating women;
* Complications require long-term immunosuppressive treatment, or systemic or local use of immunosuppressive corticosteroids (> 10mg / day prednisone or other therapeutic hormones);
* By judgment of the investigator, there are concomitant diseases that seriously endanger the safety of the patient or affect the completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
DLTs | At the end of Cycle 1 (each cycle is 28 days)
  DLTs are defined as grade 3 or higher adverse events that are related to fruquintinib during the first cycle of therapy.
RP2D | At the end of Cycle 1 (each cycle is 28 days)
  Maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D)
PFS | about 2 years
  PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first.

SECONDARY OUTCOMES:
OS | about 2 years
  The time from treatment initiation until death from any reason
ORR | about 2 years
  The proportion of patients with a confirmed complete response or partial response on two consecutive occasions≥4 weeks apart
DCR | about 2 years
  The proportion of patients with a best overall response of confirmed complete or partial response, or stable disease (CR+ PR + SD)
DoR | about 2 years
  Duration of Response is defined as the time from the first documentation of response (PR or better) to the first documented disease progression evidence (according to RECIST 1.1) of the responders
adverse events (AEs) categorized by severity in accordance with the NCI CTC AE Version 5.0 | about 2 years
  Safety and tolerance will be evaluated by incidence, severity and outcomes of adverse events (AEs) and categorized by severity in accordance with the NCI CTC AE Version 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No